CLINICAL TRIAL: NCT07392944
Title: Effects of a Multicomponent Exercise Program on Physical Function, Cognition and Falls Risk Among Older Adults Living in Nursing Homes: MOVE4CARE
Brief Title: Multicomponent Exercise Program on Physical Function, Cognition and Falls Risk Among Older Adults Living in Nursing Homes
Acronym: MOVE4CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEFADE322025
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Dementia
Keywords: Exercise; Frailty; Nursing homes; Multicomponent exercise; Falls; Cognitive function; Physical performance
MeSH Terms: conditions — Frailty; Dementia; Motor Activity | interventions — Relaxation Therapy

STUDY DESIGN:
Intervention Model Description: The study will follow a parallel, randomized clinical trial design: 12 weeks for the first intervention period, and an 18-week follow-up without any intervention.
  Data collection will occur at three time-points: baseline, 12-week (end of intervention), and 18-week follow-up (without intervention).
Who Masked: Participant, Outcomes Assessor
Masking Description: External investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent exercise (Experimental): Supervised multicomponent exercise training.
  Interventions: Other: Multicomponent exercise intervention
- stretching and relaxation program (Active Comparator): Stretches, deep breathing and relaxation exercises
  Interventions: Other: stretching and relaxation program

INTERVENTIONS:
Other: Multicomponent exercise intervention — Twice-weekly for the 12-week duration. The exercise intervention will take place at the nursing homes and consists of 12 weeks of supervised multicomponent exercise training, performed twice weekly on nonconsecutive days to avoid overtraining and fatigue. Each session will last 50-60 min and consist of a warm-up, progressive resistance and power exercises combined with aerobic and balance activities, and a 5-min cool-down period (stretching and flexibility movements). The exercise protocol will follow the Global Consensus on Optimal Exercise recommendations for enhancing healthy longevity in older adults.
  Arms: Multicomponent exercise
Other: stretching and relaxation program — Twice-weekly for the 12-week duration. The CON Program consist of stretches, deep breathing and relaxation techniques, general (light intensity) physical activity in the sitting position.
  Arms: stretching and relaxation program

SUMMARY:
Can a multicomponent exercise program significantly improve physical and cognitive function, as well as reduce falls rate in nursing home residents? To adress this question, this study aims to compare the effectiveness of a multicomponent exercose program to a stretching and relaxation program in nursing home residents.

DETAILED DESCRIPTION:
Individuals living in nursing homes often present with physical frailty and cognitive impairment. Notably, these two disabling syndromes are associated with rapid functional and cognitive decline, increased dependence, falls, hospitalization, and mortality. Long-term care requires effective interventions to promote the maintenance of functional and cognitive abilities, as well as reduce fall episodes. Non-pharmacological, particularly multicomponent exercise training has been recognized as an utmost intervention to promote health benefits among institutionalized older adults. However, findings need to be confirmed in a rigorously designed randomized controlled trial (RCT). Thus, we propose a 12-week RCT in older adults living in nursing homes to assess the efficacy of a multicomponent exercise training (resistance/power, balance and aerobic) to improve physical function, cognition and prevent falls.

Primary Question: In older adults living in nursing homes, can a multicomponent exercise program significantly improve physical and cognitive function, as well as reduce falls vs. stretching and relaxation program (i.e., active control; CON)? Secondary Questions: Do the benefits of multicomponent exercise training persist 6-week post cessation? What is the moderating role of specific subgroups (frail older adults; dementia) on the effects of multicomponent training on the outcomes of interest? Methods: A 12-week assessor-blinded, RCT, with a 6-week follow-up, in older adults living in nursing homes of Vila Nova de Gaia (Porto district), Portugal. Participants will be randomized to either: a) Multicomponent exercise training group or b) active CON. The intervention group will include 12 weeks of supervised multicomponent exercise training, performed twice weekly on nonconsecutive days to avoid overtraining and fatigue. Each session will last 50-60 min and consist of a warm-up, progressive resistance and power exercises combined with aerobic and balance activities, and a 5-min cool-down period (stretching and flexibility movements). The exercise protocol will follow the Global Consensus on Optimal Exercise recommendations for enhancing healthy longevity in older adults. The CON group will include stretches, deep breathing and relaxation techniques, general (light intensity) physical activity in the sitting position. Measurement will occur at baseline, 12, and 18 weeks, with falls tracked weekly.

ELIGIBILITY:
Inclusion Criteria:

* Ability to ambulate (with or without assistance);
* Ability to perform chair stands (with or without assistance);
* Ability to understand and properly follow testing procedures.

Exclusion Criteria:

* Any contraindication that precludes exercise performance or testing procedures, including terminal illness, uncontrolled disease, or other unstable medical conditions;
* Short Physical Performance Battery (SPPB) score < 3 points;
* Participation in any exercise intervention within the past 3 months;
* Simultaneous participation in another clinical trial during the study;
* Planned transfer to another nursing home facility, to home, or to hospitalization during the intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-18 (Estimated); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline on Short Physical Performance Battery (SPBB) | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  The Short Physical Performance Battery (SPPB) is a standardized assessment tool of lower limb function, testing 3 dimensions: standing balance, walking speed, and chair stands. Each component is scored between 0-4, total score from 0 (poor performance) to 12 (best performance).

SECONDARY OUTCOMES:
Change from Baseline on Timed Up and Go (TUG) | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  The Timed Up and Go (SPPB) is a standardized assessment of functional mobility. Briefly, the participants will be instructed to rise from a chair, walk 3 meters at their usual pace, turn around, walk back to the chair, and sit down. The time taken to complete the task was recorded and used as outcome, with longer durations representing poorer functional mobility.
Change from Baseline on Handgrip test | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  Handgrip strength will be obtained with a Digital hand dynamometer (Sammons Preston Inc., Bolingbrook, Illinois, USA). Measurements will be carried out following the American Society of Hand Therapists recommendations, and each participant will perform three attempts with a pause of 15s between trials
Falls rate | Weekly tracking over 18-week study period
  The number of self-reported falls during the 12-week intervention period (i.e., rate of falls) and follow-up (without intervention).
Change from baseline in global cognitive function as measured by the Montreal Cognitive Assessment | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  The MoCA is a brief, standardized cognitive screening tool, that enable assesses multiple cognitive domains (global cognitive function), including attention, executive functions, memory, language, visuospatial abilities, abstraction, calculation, and orientation. The test consists of a 30-point scale and typically requires approximately 10 minutes to administer. Higher scores indicate better cognitive performance.
Change from baseline in executive functions as measured by the Trail Making Test (Part A) and Digit Substitution Symbol Test | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  The Trail Making Test Part A (TMT-A) is a widely used neuropsychological measure of visual attention, processing speed, and psychomotor function. Participants are required to connect numbered circles in sequential order as quickly and accurately as possible. Performance is typically scored by completion time in seconds, with longer times indicating poorer performance. The Digit Symbol Substitution Test (DSST) is a standardized measure of processing speed, attention, working memory, and visuomotor coordination. Participants are asked to match symbols to corresponding numbers according to a reference key within a fixed time (90 seconds). The total number of correct substitutions constitutes the outcome measure, with higher scores reflecting better cognitive performance
Change from baseline in mood as measured by the Geriatric Depression Scale | Baseline, immediately after 12 weeks of intervention and after 18 weeks follow-up
  The short-version of the Geriatric Depression Scale GDS-15 is a brief, screening instrument designed to identify depressive symptoms. The total score ranges from 0 to 15, with higher scores indicating greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Joana Carvalho, PhD, Principal Investigator — Universidade do Porto
Locations (1):
- Faculty of Sports, University of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No